CLINICAL TRIAL: NCT01509105
Title: Post Marketing Surveillance To Observe Safety Of Prevenar 13
Brief Title: Prevenar13 Post Market Surveillance
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 6096A1-4029; B1851057 (Other: Alias Study Number)
Record Dates: First submitted 2011-09-30; First posted 2012-01-12 (Estimated); Results first posted 2017-02-13 (Actual); Last update posted 2017-02-13 (Actual); Status verified 2016-12

CONDITIONS: Healthy
MeSH Terms: interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group1
  Interventions: Biological: 13-valent pneumococcal vaccine

INTERVENTIONS:
Biological: 13-valent pneumococcal vaccine — 0.5mL IM (Intramuscular administration) as per recommended schedule
  Other Names: Prevenar 13

SUMMARY:
It is an observational multi-center study to assess the safety profile of Prevenar13 used among Korean children in the routine clinical setting following a licensure and introduction of the vaccine. This study is designed to fulfill regulatory requirement for any new drug authorized by KFDA.

DETAILED DESCRIPTION:
non-randomization, non-probability sampling

ELIGIBILITY:
Inclusion Criteria:

* Infants and children aged 6 weeks to 5 years, whose legally authorized representatives of patients agree to provide written informed consent form (data privacy statement).

Exclusion Criteria:

* Infants and children who are not indicated and/or contraindicated for the Prevenar13 usage will not be included.

Ages: 6 Weeks to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All infants and children meeting the usual prescribing criteria for Prevenar 13 as per the local product information for usage
Sampling Method: Non-Probability Sample
Enrollment: 649 (Actual)
Dates: Start 2011-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- South Korea (18):
  - Choi's Pediatric Clinic, Wŏnju, Gangwon-do
  - Seoul Children's Hospital, Osan, Gyeonggi-do
  - Bundang Pediatric Clinic, Seongnam-si, Gyeonggi-do
  - Teun Teun Pediatric clinic, Suwon, Gyeonggi-do
  - Namujungwon Women's Hospital, Yangju, Gyeonggi-do
  - Yonsei Pediatric Clinic, Yongin-si, Gyeonggi-do
  - Busan National University Hospital, Busan
  - Jaeil Alliance Pediatrics Clinic, Daegu
  - Teun Teun Pediatric Clinic, Daegu
  - Eulji University Hospital, Daejeon
  - Korea University Ansan Hospital, Gyeonggi-do
  - Cha Bundang Medical Center, Cha University, Gyeonggi-do
  - Inha University Hospital, Incheon
  - Lee Ha Young Pediatrics, Incheon
  - Asan Medical Center, Seoul
  - Eulji Medical Center, Seoul
  - JaMo Women's Hospital, Suyeong-gu
  - Ulsan University Hospital, Ulsan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=6096A1-4029&StudyName=Prevenar13%20post%20market%20surveillance

RESULTS

PARTICIPANT FLOW:
Groups:
- Prevenar 13: Participants aged below 6 months recieved single 0.5 milliliter (mL) dose of Prevenar 13 vaccine, intramuscularly at approximately 2, 4, 6 months of age and single 0.5 mL booster dose at least 60 days after the last dose. Participants aged between 7 to 11 months recieved 2 doses of 0.5 mL Prevenar 13 vaccine intramuscularly, at least 1 month apart and one 0.5 mL dose after the age of 12 months, separated from the previous dose by at least 2 months. Participants aged between 12 to 23 months recieved two 0.5 mL doses of Prevenar 13 vaccine intramuscularly, at least 2 months apart. Participants aged between 24 months to 17 years recieved single 0.5 mL dose of Prevenar 13 vaccine intramuscularly. Participants were followed up to 28 days after last dose of study vaccination.
Period: Overall Study
Arm/Group | Prevenar 13
Started | 649
Completed | 649
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who recieved at least 1 dose of Prevenar 13 and had the safety assessment through appropriate follow-up.
Arm/Group | Prevenar 13
Number analyzed (Participants) | 649
Age, Continuous [Mean (Standard Deviation); unit: months]
  Mean Age | 4.26 (12.86)
Gender [Count of Participants; unit: Participants]
  Female | 321
  Male | 328

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs): Within 7 Days After Vaccination 1
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. A treatment emergent AE was defined as an event that emerged during the treatment period that was absent before treatment, or worsened during the treatment period relative to the pretreatment state. AEs included both serious and non-serious adverse events.
Time Frame: Within 7 days after Vaccination 1
Population: Safety analysis set included all participants who recieved at least 1 dose of Prevenar 13 and had the safety assessment through appropriate follow-up. Here, "number of participants analyzed" (N) signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Prevenar 13
Number analyzed (Participants) | 640
participants
  Adverse Events | 68
  Serious Adverse Events | 1

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs): Within 7 Days After Vaccination 2
Description: as for outcome 1
Time Frame: Within 7 days after Vaccination 2
Population: Safety analysis set included all participants who recieved at least 1 dose of Prevenar 13 and had the safety assessment through appropriate follow-up. Here, "N" signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Prevenar 13
Number analyzed (Participants) | 536
participants
  Adverse Events | 67
  Serious Adverse Events | 0

3. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs): Within 7 Days After Vaccination 3
Description: as for outcome 1
Time Frame: Within 7 days after Vaccination 3
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Prevenar 13
Number analyzed (Participants) | 489
participants
  Adverse Events | 52
  Serious Adverse Events | 2

4. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs): Within 28 Days After Vaccination 4
Description: as for outcome 1
Time Frame: Within 28 days after Vaccination 4
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Prevenar 13
Number analyzed (Participants) | 342
participants
  Adverse Events | 43
  Serious Adverse Events | 0

5. Primary Outcome: Number of Participants With Treatment-Related Adverse Events (AEs) or Serious Adverse Events (SAEs): Within 7 Days After Vaccination 1
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Within 7 days after Vaccination 1
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Prevenar 13
Number analyzed (Participants) | 640
participants
  Adverse Events | 37
  Serious Adverse Events | 0

6. Primary Outcome: Number of Participants With Treatment-Related Adverse Events (AEs) or Serious Adverse Events (SAEs): Within 7 Days After Vaccination 2
Description: as for outcome 5
Time Frame: Within 7 days after Vaccination 2
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Prevenar 13
Number analyzed (Participants) | 536
participants
  Adverse Events | 30
  Serious Adverse Events | 0

7. Primary Outcome: Number of Participants With Treatment-Related Adverse Events (AEs) or Serious Adverse Events (SAEs): Within 7 Days After Vaccination 3
Description: as for outcome 5
Time Frame: Within 7 days after Vaccination 3
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Prevenar 13
Number analyzed (Participants) | 489
participants
  Adverse Events | 13
  Serious Adverse Events | 0

8. Primary Outcome: Number of Participants With Treatment-Related Adverse Events (AEs) or Serious Adverse Events (SAEs): Within 28 Days After Vaccination 4
Description: as for outcome 5
Time Frame: Within 28 days after Vaccination 4
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Prevenar 13
Number analyzed (Participants) | 342
participants
  Adverse Events | 17
  Serious Adverse Events | 0

9. Secondary Outcome: Duration of Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Duration of AE is the total time from onset of adverse event till the event is resolved in participants who had at least 1 AE.
Time Frame: Baseline up to 28 days after last dose of study vaccination (13 Months)
Population: Safety analysis set included all participants who recieved at least 1 dose of Prevenar 13 and had the safety assessment through appropriate follow-up. Here, "N" signifies those participants who had at least 1 adverse event.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Prevenar 13
Number analyzed (Participants) | 166
days | 7.21 (6.92)

10. Secondary Outcome: Number of Participants With Adverse Events (AEs) by Severity
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An AE was assessed according to severity; mild (not causing any significant problem, dose adjustment not required), moderate (caused problem that does not interfere significantly with usual activities or the clinical status, dose adjustment needed due to adverse event) and severe (caused problem that interferes significantly with usual activities or the clinical status, study drug stopped due to adverse event).
Time Frame: Within 7 days after Vaccination 1, 2, 3 and within 28 days after Vaccination 4
Population: Safety analysis set included all participants who recieved at least 1 dose of Prevenar 13 and had the safety assessment through appropriate follow-up. Here, "n" signifies those participants who were evaluable at specified time points.
Measure: Number; unit: participants
Arm/Group | Prevenar 13
Number analyzed (Participants) | 649
participants
  After Vaccination 1: Mild (n =640) | 66
  After Vaccination 1: Moderate (n =640) | 4
  After Vaccination 1: Severe (n =640) | 0
  After Vaccination 2: Mild (n =536) | 64
  After Vaccination 2: Moderate (n =536) | 4
  After Vaccination 2: Severe (n =536) | 0
  After Vaccination 3: Mild (n =489) | 50
  After Vaccination 3: Moderate (n =489) | 7
  After Vaccination 3: Severe (n =489) | 0
  After Vaccination 4: Mild (n =342) | 41
  After Vaccination 4: Moderate (n =342) | 2
  After Vaccination 4: Severe (n =342) | 0

11. Secondary Outcome: Number of Participants With Outcome in Response to Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Outcome of an AE was response to a question answered by those participants who had at least 1 AE: 'Is the adverse event still present?' as 'yes', 'unknown' or 'no-resolved'.
Time Frame: Baseline up to 28 days after last dose of study vaccination (13 Months)
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Prevenar 13
Number analyzed (Participants) | 166
participants
  Yes | 1
  Unknown | 1
  No-resolved | 164

12. Secondary Outcome: Number of Participants Discontinued Due to Adverse Events
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Time Frame: Baseline up to 28 days after last dose of study vaccination (13 Months)
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Prevenar 13
Number analyzed (Participants) | 649
participants | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non serious in another participant, or one participant may have experienced both a serious and non serious event during the study.
Arm/Group | Prevenar 13
Serious Adverse Events (participants affected / at risk) | 3/649
Other Adverse Events (participants affected / at risk) | 165/649
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prevenar 13 (N=649)
MEDICINE INEFFECTIVE (General disorders) | 1
PHARYNGITIS (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prevenar 13 (N=649)
INJECTION SITE RASH (Injury, poisoning and procedural complications) | 3
INJECTION SITE REACTION (Injury, poisoning and procedural complications) | 7
CRYING ABNORMAL (General disorders) | 1
FEVER (General disorders) | 40
ANOREXIA (Gastrointestinal disorders) | 1
CONSTIPATION (Gastrointestinal disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 3
ENTERITIS (Gastrointestinal disorders) | 12
GASTRO-INTESTINAL DISORDER NOS (Gastrointestinal disorders) | 2
GASTROENTERITIS (Gastrointestinal disorders) | 5
VOMITING (Gastrointestinal disorders) | 1
EAR ACHE (Ear and labyrinth disorders) | 1
LIGAMENT DISORDER (Musculoskeletal and connective tissue disorders) | 1
NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
INSOMNIA (Psychiatric disorders) | 1
NERVOUSNESS (Psychiatric disorders) | 3
ANAEMIA HYPOCHROMIC (Blood and lymphatic system disorders) | 1
BRONCHITIS (Infections and infestations) | 15
CYSTITIS (Infections and infestations) | 1
FURUNCULOSIS (Infections and infestations) | 1
INFECTION VIRAL (Infections and infestations) | 1
OTITIS MEDIA (Infections and infestations) | 7
PHARYNGITIS (Infections and infestations) | 33
PNEUMONIA (Infections and infestations) | 11
PYELONEPHRITIS (Infections and infestations) | 2
RHINITIS (Infections and infestations) | 19
SINUSITIS (Infections and infestations) | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 38
COUGHING (Respiratory, thoracic and mediastinal disorders) | 11
SPUTUM DISORDER (Respiratory, thoracic and mediastinal disorders) | 3
DERMATITIS (Skin and subcutaneous tissue disorders) | 7
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 2
ECZEMA (Skin and subcutaneous tissue disorders) | 6
PRURITUS (Skin and subcutaneous tissue disorders) | 1
RASH (Skin and subcutaneous tissue disorders) | 3
SEBORRHOEA (Skin and subcutaneous tissue disorders) | 1
SKIN DISORDER (Skin and subcutaneous tissue disorders) | 4
URTICARIA (Skin and subcutaneous tissue disorders) | 3
CONJUNCTIVITIS (Eye disorders) | 1
HETEROPHORIA (Eye disorders) | 1
LACRIMAL DUCT OBSTRUCTION (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.